CLINICAL TRIAL: NCT00670943
Title: Effect of Abrupt Plavix® Discontinuation on Platelet Function
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Collaborators: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Jean G. Diodati, Hôpital du Sacré-Coeur de Montréal
Other Study IDs: C.E. 2007-05-41
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel discontinuation; Platelet aggregation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Patients with stable CAD with scheduled discontinuation of clopidogrel
  Interventions: Other: Platelet function testing
- B: Patients with stable CAD not taking clopidogrel
  Interventions: Other: Platelet function testing

INTERVENTIONS:
Other: Platelet function testing

SUMMARY:
The well established importance of regular administration of antiplatelet drugs stands on firm grounds, as large meta-analyses have shown these therapies to significantly reduce the risk of death. Plavix® (clopidogrel) is widely used following coronary angioplasty, to reduce the risk of periprocedural thrombotic complications, for up to one year. As the current recommendations suggest clopidogrel use for no longer than one year, the drug is normally discontinued within that period. In the limited state of knowledge on antiplatelet drug withdrawal, an early sound of alarm has risen from early thromboembolic complications reported after the interruption of antiplatelet treatment used in prevention of ischemic vascular disease. Although little information is available, discontinuation of thienopyridines has been associated with increased thromboembolic complications, mainly acute stent thrombosis. These complications may signal a platelet sensitization effect to aggregating stimuli by antiplatelet drugs taken chronically.

The current study aims to evaluate the impact of clopidogrel discontinuation on platelet function, in order to shed light on underlying mechanisms leading to increased risk of acute thrombo-occlusive events.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Patients suffering from stable CAD scheduled to discontinue clopidogrel therapy at least one month after stent implantation
* Group 2: Stable clopidogrel-naïve CAD patients
* Patients willing to participate in the study and to sign the informed consent form

Exclusion Criteria:

* Acute coronary syndrome or revascularization in the last 3 months prior to enrolment
* Concurrent ingestion of nonsteroidal anti-inflammatory drugs (NSAIDs, including COX-2 selective anti-inflammatory drugs), ticlopidine, dipyridamole, warfarin or acenocoumarol
* Major surgical procedure within 1 month before enrolment
* Platelet count outside the 100 000 to 450 000/μL range
* Hematocrit < 25% or haemoglobin < 100 g/L
* Patient undergoing dialysis for chronic renal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Diodati, MD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada